CLINICAL TRIAL: NCT04173260
Title: The AUDYT Trial: An Open-label Study to Define the Safety, Tolerability and Clinical Activity of Deutetrabenazine (AUstedo) in Adult Study Subjects With DYsTonia
Brief Title: An Open-label Study to Define the Safety, Tolerability and Clinical Activity of Deutetrabenazine (AUstedo) in Adult Study Subjects With DYsTonia
Acronym: AUDYT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10070487
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Dystonia, Primary
MeSH Terms: conditions — Dystonic Disorders | interventions — deutetrabenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention arm - Oral Deutetrabenazine (Experimental): This is the only arm for this trial. All subjects will receive oral Deutetrabanazine.
  Interventions: Drug: Deutetrabenazine 6 MG

INTERVENTIONS:
Drug: Deutetrabenazine 6 MG — Increasing doses of Deutetrabenazine

SUMMARY:
This is a single-center, open-label study of AUSTEDO in study subjects with dystonia. The study will provide preliminary experience of the safety, tolerability, and clinical activity of AUSTEDO in study subjects with dystonia. Study duration will be up to 13 weeks from screening (Visit 1) to the post treatment evaluation (Visit 5). Treatment period from drug initiation to final on-treatment Visit will be 12 weeks, or less, as follows: during the ramp-up period, study drug will start at 12 mg/day (6 mg twice daily) and will be titrated weekly by 6 mg/day increments until either 1) the maximal allowable dose (48 mg/day) is reached, or 2) dose-limiting side-effects occur. In study subjects receiving a strong CYP2D6 inhibitor, the maximum allowed dose of AUSTEDO will be 36 mg/day, reducing study duration (due to a reduction in the ramp-up period) to 11 weeks. Study subjects who experience dose-limiting side effects will be maintained on their maximum tolerated dose. Once the maximal dose is established for each participant, they will complete 6 continuous weeks on this dose (maintenance period), followed by a 1-week washout. For study subjects unable to titrate up to 48 mg/day due to side effects, the 6 weeks of maintenance will start once they reduce the study drug back to the maximum well-tolerated dose. Adverse events will be monitored throughout the study and will be reported after drug initiation. Dose reductions, suspensions, and withdrawals due to adverse events will be recorded. ECG readings will be measured at screening, during week 2, during the first week of the maintenance period (whenever this is established to be, typically week 7 for subjects able to titrate up to 48 mg/day), immediately before washout (week 12 for those study subjects who are able to titrate up to 48 mg/day) and during week 13. Assessment of Columbia Suicide Severity Rating Scale and Epworth Sleepiness Scale scores will occur at screening and all clinic Visits. The Mini Mental (MMSE) Scale will be performed at screening and at the final on-treatment Visit (week 12). A video examination of the study subjects will be made at screening (right before initiation of the study drug), and after 6 weeks on AUSTEDO at a steady dose (right before drug cessation). Part III of the MDS-UPDRS will be performed at both of these Visits as well to screen for the appearance of drug-induced parkinsonism. Videos will be sent to raters blinded to treatment, Visit number and recording date.

ELIGIBILITY:
Inclusion Criteria:

1. Study subjects with definite dystonia, as established by a movement disorder specialist.
2. Study subjects of any race and either gender, age 18 or more on the date the informed consent form (ICF) is signed and with the capacity to provide voluntary informed consent.
3. Study subjects able to read and understand English and the ICF and are willing to comply with all study procedures, treatment and follow-up.
4. Study subjects who are taking any central nervous system acting medications (e.g., benzodiazepines, antidepressants, hypnotics), including medications for the treatment of dystonia, will be on a stable regimen for at least 30 days prior to the screening Visit, and will willing to remain on the same dose for the duration of the study.
5. Female of child-bearing potential will not be pregnant and will be using an acceptable method of contraception.
6. Study subjects with an MMSE >24.

Exclusion Criteria:

1. Exposure to dopamine blockers prior to the onset of dystonia that could, in the investigator's opinion, have caused dystonia.
2. Study subjects with genetically-confirmed dopa-responsive dystonia.
3. Study subjects with a diagnosis of Parkinson's or an atypical parkinsonian syndrome.
4. Study subjects with a history of bipolar disorder or major depression, or the presence of active depression.
5. Study subjects with a history of a suicide attempt or suicidal ideations, as well as the presence of active suicidal ideation as detailed on the C-SSRS administered during Visit 1.
6. Study subjects with a history of schizophrenia or schizophrenia spectrum disorders.
7. Treatment with tetrabenazine, reserpine, valbenazine, a monoamino oxidase inhibitor, a-methyl-p-tyrosine, strong anticholinergic medications, metoclopramide, antipsychotics, dopamine agonists, levodopa, and/or stimulants within 30 days of screening.
8. Treatment with botulinum toxin less than 11 weeks prior to screening (Visit 1); subjects receiving injections sooner than every 12 weeks will be excluded if their next injection is scheduled farther than 6 days from screening.
9. Presence of a neurologic condition that could confound dystonia assessments.
10. Study subjects with a history of clinically relevant hepatic disease.
11. Study subjects with a history of renal insufficiency.
12. Any unstable medical illness.
13. A corrected QT (Bazett) interval of 450 (458) milliseconds in men or 460 (472) milliseconds in women on 12-lead ECG at screening, or a history of cardiac arrhythmias.
14. Study subjects participating in any drug or device clinical investigation concurrently or within 30 days prior to screening for this study.
15. Study subjects with a known hypersensitivity or contraindication to the study drug or its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifteen subjects were recruited between April 2021 and December 2023.
Pre-assignment Details: All subjects received IP; there was no placebo arm.
Period: Overall Study
Arm/Group | Intervention Arm - Oral Deutetrabenazine
Started | 15
Completed | 11
Not Completed | 4
Not completed — Early termination | 4

BASELINE CHARACTERISTICS:
Population: Adults with non-dopa responsive isolated dystonia
Arm/Group | Intervention Arm - Oral Deutetrabenazine
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 63 [29 to 74]
Sex: Female, Male [Count of Participants; unit: Participants] — The variable "sex" referred to sex assigned at birth, self reported.
  Participants
    Female | 11
    Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Study Subjects Able to Titrate up to the Maximum Tolerated Dose
Description: Proportion of study subjects able to titrate up to 48 mg/d (or up to 36 mg/d if receiving a strong CYP2D6 inhibitor) and able to complete the study at this dosage
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Arm - Oral Deutetrabenazine: All subjects in this study received IP in an open label fashion
Arm/Group | Intervention Arm - Oral Deutetrabenazine
Number analyzed (Participants) | 15
Participants | 6

2. Secondary Outcome: Number of Participants With Change in Suicidality
Description: Documentation of change in the Columbia Suicide Severity Rating Scale. Items on this scale are both binary (Yes/No) and numeric (0-5). "No" answers and lower numeric values indicate a better outcome.
Time Frame: Baseline and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm - Oral Deutetrabenazine
Number analyzed (Participants) | 15
Participants | 0

3. Secondary Outcome: Change in Median Daytime Somnolence Score Among Subjects
Description: Documentation of change in the Stanford Sleepiness Scale. Scale was assessed at the initial and last study visit; difference was calculated between both scores, and reported herein as a median among all participants' scores and full range.
  Items on this scale are numeric (1-7). Lower numeric values indicate a better outcome.
Time Frame: Baseline and 3 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Arm - Oral Deutetrabenazine
Number analyzed (Participants) | 15
score on a scale | 0 [-5 to 2]

4. Secondary Outcome: Change in Median MMSE Score Among Subjects
Description: Documentation of change in the Mini Mental Scale. Scale was assessed at the initial and last study visit; difference was calculated between both scores, and reported herein as a median among all participants' scores and full range.
  The higher the total score on this scale, the better the outcome. Values range from 0 to a maximum of 30.
Time Frame: Baseline and 3 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Arm - Oral Deutetrabenazine
Number analyzed (Participants) | 15
score on a scale | 1 [-4 to 3]

5. Secondary Outcome: Development of Parkinsonism, as Determined by Change in Median MDS-UPDRS III Score Among Subjects
Description: Documentation of change in the MDS-Unified Parkinson's Disease Rating Scale, Part III. Scale was assessed at the initial and last study visit; difference was calculated between both scores, and reported herein as a median among all participants' scores and full range.
  The lower the total score on this scale, the better the outcome. Values range from 0 to a maximum of 128.
Time Frame: Baseline and 3 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Arm - Oral Deutetrabenazine
Number analyzed (Participants) | 15
score on a scale | 2 [-19 to 13]

6. Secondary Outcome: Change in Median PGI-I Score
Description: Documentation of change in the Patient Global Impression of Improvement Scale (PGI-I). This is a Likert scale, with values from 1-7. A value of 1 indicates the best outcome. A value of 4 indicates no perceived change.
Time Frame: Baseline and 3 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Arm - Oral Deutetrabenazine
Number analyzed (Participants) | 15
score on a scale | 4 [1 to 5]

7. Secondary Outcome: Change in Dystonia Severity, as Determined by the Change in Median GDS Score
Description: Documentation of change in the Global Dystonia Rating Scale. Scale was assessed blindly from videos captured at the initial and last study visit; difference was calculated between both scores, and reported herein as a median among all participants' scores and full range.
  The lower the total score on this scale, the better the outcome. Values range from 0 to a maximum of 140.
Time Frame: Baseline and 3 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Arm - Oral Deutetrabenazine
Number analyzed (Participants) | 15
score on a scale | 0 [-12 to 2]

ADVERSE EVENTS:
Time Frame: Up to 13 weeks
Arm/Group | Intervention Arm - Oral Deutetrabenazine
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm - Oral Deutetrabenazine (N=15)
Suicidal depression (Psychiatric disorders) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm - Oral Deutetrabenazine (N=15)
Fatigue (Nervous system disorders) | 6
Somnolence (Nervous system disorders) | 3
COVID-19 infection (Respiratory, thoracic and mediastinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 1
Akathisia (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
* Open label design
* Patients were allowed to continue receiving BoNT injections during the trial
* No genetic testing pursued
* Patients with different phenomenologies were allowed to participate and data analyzed in aggregate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT04173260/Prot_SAP_002.pdf
  • Informed Consent Form (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT04173260/ICF_003.pdf